CLINICAL TRIAL: NCT06446024
Title: Post Market Surveillance to Evaluate the Efficacy and Safety of the INDIGO Aspiration System in Japan
Acronym: JapanIndigoPMS
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 27548
Record Dates: First submitted 2024-05-13; First posted 2024-06-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Acute Limb Ischemia; Arterial Occlusion Mesenteric Artery Superior; Acute DVT of Lower Extremity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Group 1: Indigo Aspiration System treatment: Mechanical aspiration thrombectomy
  Interventions: Device: Mechanical aspiration thrombectomy

INTERVENTIONS:
Device: Mechanical aspiration thrombectomy — Mechanical thrombectomy is an endovascular technique for removing blood clots from vessels. Penumbra's Indigo system actively extracts thrombus using a continuous vacuum pump, enabling aspiration of thrombus of various sizes and lengths.

SUMMARY:
This study aims to confirm the safety and effectiveness of the INDIGO Aspiration System in patients requiring immediate treatment for acute lower extremity artery occlusion, acute superior mesenteric artery occlusion, or severe acute deep vein thrombosis. Primary objective of the study is to collect predetermined data on use, safety and effectiveness, including clinical and technical performance of the INDIGO System in Japan.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet Appropriate Use Criteria per local Japanese requirements for acute lower limb artery, acute upper mesentery artery occlusions, or severe acute deep vein thrombosis.

Exclusion Criteria:

Patients who do not meet Appropriate Use Criteria per local Japanese requirements for acute lower limb artery, acute upper mesentery artery occlusions, or severe acute deep vein thrombosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The INDIGO System is intended for use in patients with acute lower limb artery occlusion, acute superior mesenteric artery occlusion, or severe acute deep vein thrombosis who require immediate treatment and for whom it is difficult to perform surgical thrombectomy or who are expected to have no effective therapeutic effect.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
ALI: Target Limb Salvage | 30 days post-treatment and 6 months post-treatment
  Target lower extremity salvage rate at (defined as: freedom from major amputation at or proximal to the ankle)
ALI: Technical Success | Intraoperative
  Primary technical success should be defined per vessel treated on an intent-to-treat basis and applies only to segment treated with Indigo. Defined as successful use of the device to re-establish any antegrade flow and complete or near complete (95% by volume) removal of thrombus as assessed by visual analysis of angiographic images or by other objective imaging such as DUS, CTA, or MRA.
ALI: Major device-related bleeding in ALI patients | Periprocedural
  Major bleeding events as defined by ISTH
SMA: Technical success | Intraoperative
  Restoration of antegrade blood flow without the need for other revascularization procedures such as vascular surgery or bypass.
SMA: Device-related Distal Embolization | Intraoperative
  A distal filling defect with an abrupt cut-off, determined to be new since the pre-procedure angiogram, present at the end of the procedure, and clinically significant requiring intervention other than Indigo use. If the area in question was not clearly visualized, filling defects distal to the target lesion cannot be categorized as emboli.
DVT: Technical success | Intraoperative
  Complete or near complete (75% or more) reduction in venous thrombosis, as assessed by visual evaluation of intraoperative venography
DVT: Major Device-Related Bleeding | Periprocedural
  Major device-related bleeding as defined by ISTH
DVT: New Symptomatic Pulmonary Embolism (PE) | 30 days post-treatment
  Symptomatic new PE objectively confirmed on Computed Tomographic Pulmonary Angiography (CTPA), echocardiography, MRI, or invasive contrast pulmonary angiography.
DVT: Clinically significant re-thrombosis of the target venous segment | 30 days post-treatment
  Re-thrombosis of target vein segment requiring re-intervention within 30 days
All Disease States: Device-related Serious adverse effects (SAE) and mortality | 6 months post-treatment
  Device related SAE and all-cause mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Nara City Hospital, Nara, Japan

IPD SHARING:
Plan to Share IPD: No